CLINICAL TRIAL: NCT02001350
Title: Carotid Ultrasound Study
Status: Completed | Type: Observational
Sponsor: Noblewell (Industry)
Collaborators: Cibiem, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CIB-USG.GDA.PL
Record Dates: First submitted 2013-11-22; First posted 2013-12-04 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Resistant Hypertension
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Resistant hypertension
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography

SUMMARY:
To use carotid ultrasound to screen 20-30 patients with longstanding or resistant hypertension for carotid atherosclerotic disease and bifurcation anatomy. This will establish a screening protocol for Cibiem's eventual endovascular carotid body modulation trial and will give insight into the prevalence and specific location of carotid plaque at the bifurcation in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Uncontrolled hypertension on 3 or more medications or longstanding controlled hypertension on 4 or more medications.

Exclusion Criteria:

* Previous stroke
* Carotid endarterectomy or carotid stent procedure
* >50% stenosis anywhere in carotid arteries

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients with longstanding or resistant hypertension
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Specific location of carotid plaque at the bifurcation | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paul A. Sobotka, MD, Study Director — Cibiem, Inc.
Locations (1):
- Department of Hypertension and Diabetology, Medical University of Gdansk, Gdansk, Poland